CLINICAL TRIAL: NCT05327712
Title: Using Emails and Personalized Phone Calls to Increase Affordable Care Act Marketplace Enrollment Among Households Losing Medicaid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Office of Evaluation Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Andrew Feher, Research Scientist, Office of Evaluation Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 042022
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Health Behavior
Keywords: Affordable Care Act; randomized controlled trial; Medicaid
MeSH Terms: conditions — Health Behavior | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Experimental): The control group was assigned to receive no outreach beyond an initial eligibility determination notice
  Interventions: Behavioral: Control group
- Email-only (Experimental): An email-only group assigned to receive an initial eligibility determination plus email reminders about signing up for marketplace coverage
  Interventions: Behavioral: Email only
- Phone-only (Experimental): A phone-only group assigned to receive an initial eligibility determination plus a phone call offering enrollment assistance from a service center representative (SCR);
  Interventions: Behavioral: Phone only
- Phone and email (Experimental): A phone + email group assigned to receive an initial eligibility determination, email reminders about signing up for marketplace coverage and a phone call offering enrollment assistance.
  Interventions: Behavioral: Phone and email

INTERVENTIONS:
Behavioral: Control group — No outreach during the intervention period beyond an initial eligibility notice.
  Other Names: No outreach
  Arms: Control
Behavioral: Email only — Email reminders in addition to an initial eligibility notice.
  Arms: Email-only
Behavioral: Phone only — Phone call offering enrollment assistance in addition to an initial eligibility notice.
  Arms: Phone-only
Behavioral: Phone and email — Phone call and email reminders in addition to an initial eligibility notice.
  Arms: Phone and email

SUMMARY:
Since its passage in 2010, the Affordable Care Act (ACA) has helped reduce the uninsured rate to record lows, but changes in insurance coverage over time, known as churn, remain a concern. A recent survey found that nearly 25 percent of respondents reported a change in coverage over the previous twelve months. Among the most common reasons for churn is the loss of Medicaid eligibility, placing low-income populations at risk of a coverage gap. To date, little evidence exists on effective strategies states can use to facilitate Medicaid to Marketplace coverage transitions, an issue that has become more pressing amid projections that upwards of 15 million people could lose Medicaid eligibility once the COVID-19 public health emergency expires.

To address this gap and to inform Marketplace administrators, during a Special Enrollment Period (SEP) in 2017 in California's ACA Marketplace, we conducted a randomized controlled trial to examine the effect of email reminders, personalized telephone outreach, as well as the combination of the two forms of outreach on ACA enrollment among households who recently lost Medicaid and became eligible for subsidized Marketplace coverage.

During the SEP at the end of August 2017, the investigators randomly assigned households to one of four arms based on the last digit of their household identifier: a control group assigned to receive no outreach beyond an initial eligibility determination notice; an email-only group assigned to receive an initial eligibility determination plus email reminders about signing up for marketplace coverage; a phone-only group assigned to receive an initial eligibility determination plus a phone call offering enrollment assistance from a service center representative (SCR); a phone + email group assigned to receive an initial eligibility determination, email reminders about signing up for marketplace coverage and a phone call offering enrollment assistance.

ELIGIBILITY:
Inclusion Criteria:

* Those who recently lost Medicaid eligibility and became eligible for subsidized Affordable Care Act coverage

Exclusion Criteria:

* Those who recently lost Medicaid eligibility and were found ineligible for subsidies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2173 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
Percent of households enrolled in an ACA plan by the end of the October 2017 | Two months
  Percent of households enrolled in an ACA plan during the intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Feher, PhD, Principal Investigator — Covered California
Locations (1):
- Covered California, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers are committed to sharing as much data as possible for replication, consistent with the privacy and security requirements of the state agency that govern the re-disclosure of the data.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will be available with investigator support upon publication.
Access Criteria: Replication data can be accessed via request to the primary investigator upon publication.

REFERENCES:
- [Derived] Ravel K, Ahrary J, Avakian K, Feher A, Menashe I. Effect of Personalized Outreach on Medicaid to Marketplace Coverage Transitions: A Randomized Clinical Trial. JAMA Health Forum. 2022 Oct 7;3(10):e223616. doi: 10.1001/jamahealthforum.2022.3616. PMID 36239955